CLINICAL TRIAL: NCT03004820
Title: Feasibility of Applying Remote Ischemic Conditioning in Secondary Prevention in Patients With Minor Ischemic Stroke or Transient Ischemic Attack -A Single-arm Futility Study
Brief Title: Prevention of Ischemic Conditions in Non-disabling Stroke/Transient Ischemic Attack With Remote Ischemic Conditioning
Acronym: PICNIC-ONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming, Professor, Chief Surgeon, Vice President, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RICMIS/TIA
Record Dates: First submitted 2016-12-10; First posted 2016-12-29 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Transient Ischemic Attack; Non-disabling Stroke
Keywords: Minor Ischemic Stroke; Transient Ischemic Attack; Remote Ischemic Conditioning
MeSH Terms: conditions — Ischemic Attack, Transient

STUDY DESIGN:
Intervention Model Description: Patients will receive remote ischemic conditioning
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Remote Ischemic Conditioning (Experimental): RIC (remote ischemic conditioning) consists of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on bilateral upper limbs twice a day. Medication strategy is based on physician's best judgement.
  Interventions: Device: Remote Ischemic Conditioning

INTERVENTIONS:
Device: Remote Ischemic Conditioning — RIC consist of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on bilateral upper limbs twice a day. Medication strategy is based on physician's best judgement.

SUMMARY:
This is a single-arm, open-labeled and phase II futility study. Application of Remote ischemic conditioning (RIC) as an adjunctive therapy to medication were involved in the study. The study is to test whether RIC is effective in preventing ischemic evens after a minor ischemic stroke/transient ischemic attack within 3 months and to explore the safety and compliance of chronic RIC. Medication strategy is based on physician's best judgement.

DETAILED DESCRIPTION:
This is a single-arm, open-labeled and phase II futility study. Application of Remote ischemic conditioning (RIC) as an adjunctive therapy to medication were involved in the study. RIC consisted of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on bilateral upper limbs twice a day. The study is to test whether RIC is effective in preventing ischemic evens after a minor ischemic stroke/transient ischemic attack within 3 months and to explore the safety and compliance of chronic RIC. Medication strategy is based on physician's best judgement.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years old or older of any gender or race;
2. Diagnosed with a non-cardiogenic MIS/TIA within 14 days; MIS is defined by an ischemic stroke of score of 3 or less on the NIHSS at the time of inclusion, TIA is defined as neurologic deficit attributed to focal brain ischemia, with symptoms resolution within 24 h of symptom onset, Symptom onset is defined by the "last see normal" principle;
3. Stable vital signs, normal cardiac, hepatic and renal functions;
4. Able to consent by himself/herself or by legally authorized representative.

Exclusion Criteria:

1. Diagnosis of hemorrhage or other pathology, such as vascular malformation, tumor, abscess or other non-vascular diseases, based on brain CT or MRI;
2. Modified Rankin Scale score > 2 at inclusion;
3. Received iv. recombinant tissue plasminogen activator (rtPA) therapy or interventional treatment for the current event;
4. Contradiction for aspirin or clopidogrel (known allergy, severe asthma or heart failure et al.) ;
5. Clear indication for anticoagulation therapy ( cardiac source of embolus);
6. Hemorrhagic tendency of any reason （including but not limit to Hemostatic disorder, platelet count <100 × 109/L, history of drug-induced hepatic dysfunction）;
7. Any hemorrhagic transformation;
8. Gastrointestinal bleed or major surgery within 3 months of symptoms onset;
9. Stroke or TIA induced by interventional therapy or surgery;
10. Any upper extremity soft tissue, vascular injury or peripheral blood vessel disease which may contraindicate RIC;
11. Systolic blood pressure greater than 200 mmHg after medication;
12. Planned revascularization (any angioplasty or vascular surgery) within the next 3 months ；
13. Scheduled for surgery or interventional treatment requiring RIC cessation within next 3 months;
14. Severe noncardiovascular comorbidity with life expectancy < 3 months;
15. Pregnancy;
16. Currently receiving an investigational drug or device by other studies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Recurrent rate of ischemic stroke/transient ischemic stroke | within 3 months

SECONDARY OUTCOMES:
Treatment-Related Adverse Events | within 3 months
  pain and tolerability, redness, bleeding, palpitation
Compliance of remote ischemic conditioning | within 3 months
  the proportion of patients fulfill the treatment
Incidence rate of vascular events | within 3 months
  hemorrhage stroke, myocardial infarction and vascular death
Improvements in NIH Stroke Scale | within1, 3 months
  improvements in NIH Stroke Scale in patients without recurrence or vascular events
Improvements in modified Rankin Scale | within 1, 3 months
  improvements in modified Rankin Scale Scale in patients without recurrence or vascular events
Improvements in Barthel Scale | within 1,3 months
  improvements in Barthel Scale in patients without recurrence or vascular events

OTHER OUTCOMES:
Recurrent rate of ischemic stroke/transient ischemic stroke within 1 months | within 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD, PhD, Principal Investigator — Xuanwu Hospital, Beijing; Wuwei Feng, MD, MS, Study Director — Medical University of South Carolina
Locations (4):
- China (4):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Taoyuan People's Hospital, Changde, Hunan
  - Shengli Oilfield Center Hospital, Dongying, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu SM, Zhao WL, Song HQ, Meng R, Li SJ, Ren CH, Ovbiagele B, Ji XM, Feng WW. Rationale and Study Design for a Single-Arm Phase IIa Study Investigating Feasibility of Preventing Ischemic Cerebrovascular Events in High-Risk Patients with Acute Non-disabling Ischemic Cerebrovascular Events Using Remote Ischemic Conditioning. Chin Med J (Engl). 2018 Feb 5;131(3):347-351. doi: 10.4103/0366-6999.223849. PMID 29363651